CLINICAL TRIAL: NCT06960525
Title: Comparison of Joint Mobilization vs. Strengthening Exercises for Improving Cervical Proprioception in Individuals With Nonspecific Neck Pain: A Randomized Clinical Trial
Brief Title: Joint Mobilization vs. Strengthening Exercises on Cervical Proprioception for Nonspecific Neck Pain
Acronym: CervPro-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: Al Hada Military Hospital (Other)
Responsible Party: Principal Investigator, Faisal Fahad Alharthi, Principal investigator, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-PGS-2024-03-574; 14-2024-06-07-95 (Registry Identifier: CREC- MODHS /NCBE-KACST)
Record Dates: First submitted 2025-04-06; First posted 2025-05-07 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-05

CONDITIONS: Chronic Neck Pain; Nonspecific Neck Pain
Keywords: chronic neck pain; Nonspecific neck pain; cervical proprioception; cervical mobilization; cervical strengthening exercises; neck; cervical; proprioception; mobilization; manual; strengthening; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a double-blinded randomized clinical trial with a parallel-group design.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint mobilization group (Experimental): This group will receive passive cervical joint mobilization following Maitland's approach for 3 sets of 1 minute on the most painful segment with one minute rest between sets. The specific technique and most painful level will be determined during the clinical examination. The participant lies prone on a treatment bed, then the therapist uses both thumbs to apply grade III or IV based on the patient's irritability using posteroanterior pressure to the cervical spinous process or articular pillar, with a rhythm of 2 to 3 Hz per second. This intervention could be applied in different positions of the cervical spine, depending on the patient's response, in a pain-free manner.
  Interventions: Other: Cervical joint mobilization
- Strengthening exercises group (Experimental): The exercise program will include concentric and eccentric training of the craniocervical, cervical flexors, extensors, muscles involved in cervical spine rotation and axioscapular muscles. The strengthening exercises with high frequency - low intensity will be performed. Low frequency - high intensity will be implemented when the patient's irritability is low.
  Interventions: Other: cervical strengthening exercises

INTERVENTIONS:
Other: Cervical joint mobilization — Passive cervical joint mobilization following Maitland's approach for 3 sets of 1 minute on the most painful segment with one minute rest between sets.
  Arms: Joint mobilization group
Other: cervical strengthening exercises — concentric and eccentric training of the craniocervical, cervical flexors, extensors, muscles involved in cervical spine rotation and axioscapular muscles.
  Arms: Strengthening exercises group

SUMMARY:
This clinical trial aims to compare the effects of cervical joint mobilization versus cervical strengthening exercises in patients with chronic neck pain. The study will assess neck proprioception, pain intensity, cervical muscle strength, range of motion, and neck disability.

The main question it aims to answer is:

Which treatment is superior, or do they have equal effects after the first session and after the 12th session?

Participants will:

Receive either cervical joint mobilization or cervical strengthening exercises for 12 sessions.

Do not perform any physical therapy treatment outside the trial. Visit the clinic three times per week for treatment.

DETAILED DESCRIPTION:
Neck pain refers to a type of generalized neck discomfort characterized by mechanical features. This condition is a widespread issue, causing significant levels of pain, disability, and can lead to economical strain. Patients suffering from neck pain often experience functional impairments, including weak neck muscles and impaired proprioception. Strengthening exercises and cervical joint mobilization offer effective relief of pain and improve disability. Exploring the superiority of these techniques in improving cervical proprioception to prevent recurrence is still a vague topic. Therefore, this study will investigate the effect of Maitland joint mobilization versus cervical strengthening exercises in patients with nonspecific chronic neck pain on neck proprioception, pain intensity, cervical muscles strength, range of motion and neck disability. This is a double-blinded randomized clinical trial with a parallel-group design. Twenty-six participants will be allocated randomly to one of two groups. Group one (Mobilization) will have cervical joint mobilization according to Maitland approach. Group two (Exercises) will perform craniocervical, cervical and axioscapular muscles strengthening exercises. Treatment will be provided for 12 sessions. Both groups will receive standardized care, including patient education and transcutaneous electrical nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years
* Pain ≥ 3 months
* Neck pain on VAS ≥ 3/10
* NDI ≥ 5/50 points
* ZZ Errors ≥ 9 or the time to complete the task ≥ 28s

Exclusion Criteria:

* Unilateral headache aggravated by neck movement.
* Upper extremity symptoms beyond the elbow.
* Any history of neck trauma including whiplash
* Recent fractures (last 8 weeks)
* Cervical surgery (last 3 months)
* Current neck-related dizziness
* Known or suspected ves3bular pathology
* Internal fixation of the cervical spine
* Physical therapy for the neck (last 3 months)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Active cervical movement sense | Three points: 1) baseline, 2) immediately after intervention, and 3) week 4
  Participants will be comfortably seated upright on a chair with a backrest, positioned 1 meter away from a board displaying a zigzag pattern (ZZ). They will wear a headband with a laser pointer attached. The pattern is affixed to the board in a manner that directs the laser beam to the pattern's centre.
Cervical joint position error | Three points: 1) baseline, 2) immediately after intervention, and 3) week 4
  Participants were comfortably seated upright on a chair with a backrest, positioned 0.9 meters away from a wall. Using a distance laser meter, for accurate measurement, the distance between the forehead of the participant and the wall was measured after the participant wore a headband with a laser pointer attached. A point on the wall was located as the patient was in a self-neutral position. A warm-up session was given as the patient with open eyes was instructed to perform flexion, extension, and rotation on both sides and return to the selected point after each movement. After that, the patient was asked to perform the movement for three trials in each movement direction with their eyes closed.

SECONDARY OUTCOMES:
Visual Analogue Scale | Three points: 1) baseline, 2) immediately after intervention, and 3) week 4
  Pain intensity was assessed using the Visual Analogue Scale (VAS) which a ruler with 100 mm measured. The 0 mm indicates 'No pain" and 100 mm indicates " worse pain". Patient were asked to mark their level of pain.
Cervical muscles strength | Three points: 1) baseline, 2) immediately after intervention, and 3) week 4
  Measure the cervical muscles using a hand-held dynamometer. The patient was asked to perform flexion, extension, lateral flexion and rotation to both sides.
Cervical range of motion | Three points: 1) baseline, 2) immediately after intervention, and 3) week 4
  The range of motion was measured three times in flexion, extension, left-right lateral flexion and rotation using a therapeutic range of motion inclinometer.
Neck Disability Index | Three points: 1) baseline, 2) week 4
  Neck Disability Index (NDI) was used to evaluate the score of self-rated disability linked to neck pain experienced during the preceding week. This assessment consists of 10 questions, each question rated from 0 (indicating no disability) to 5 (representing total disability), with a maximum score of 50 points (see Appendix D.). Disability can be categorized as no disability (0-4 points), mild disability (5-14 points), moderate disability (15-24 points), severe disability (25-34 points), and (35-50 points) present complete disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ali M Alshami, Phd, Study Director — Imam Abdulrahman Bin Faisal University
Locations (1):
- Armed Forces Hospital - Al Hada, Ta'if, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] de Zoete RMJ. Exercise Therapy for Chronic Neck Pain: Tailoring Person-Centred Approaches within Contemporary Management. J Clin Med. 2023 Nov 15;12(22):7108. doi: 10.3390/jcm12227108. PMID 38002720
- [Background] de Zoete RM, Armfield NR, McAuley JH, Chen K, Sterling M. Comparative effectiveness of physical exercise interventions for chronic non-specific neck pain: a systematic review with network meta-analysis of 40 randomised controlled trials. Br J Sports Med. 2020 Nov 2:bjsports-2020-102664. doi: 10.1136/bjsports-2020-102664. Online ahead of print. PMID 33139256
- [Background] Ernst MJ, Williams L, Werner IM, Crawford RJ, Treleaven J. Clinical assessment of cervical movement sense in those with neck pain compared to asymptomatic individuals. Musculoskelet Sci Pract. 2019 Oct;43:64-69. doi: 10.1016/j.msksp.2019.06.006. Epub 2019 Jul 2. PMID 31277033